CLINICAL TRIAL: NCT07322822
Title: Effectiveness of an Active Coping Program on Pain, Disability, and Psychosocial Factors in Patients With Chronic Musculoskeletal Pain: A Controlled Clinical Study
Brief Title: Active Coping Program for Chronic Musculoskeletal Pain: A Controlled Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Clinical Professor, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11
Record Dates: First submitted 2025-12-16; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Chronic Musculoskeletal Pain; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Coping Program (Experimental)
  Interventions: Behavioral: Active Coping Program
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Active Coping Program — Participants assigned to this arm will receive an 8-week active coping program for chronic musculoskeletal pain. The program is a multimodal, non-pharmacological intervention aimed at improving self-management and active pain coping. Core components include pain education (e.g., understanding chronic pain mechanisms), movement-based therapeutic exercise/graded activity, and behavioral strategies to address maladaptive pain-related beliefs and behaviors (e.g., fear of movement and pain catastrophizing). The intervention is delivered following a standardized protocol to ensure consistency across participants.
  Arms: Active Coping Program
Other: Usual Care — Participants assigned to this arm will receive usual care as provided in routine clinical practice in primary care. No additional study-specific intervention is delivered. Usual care may include standard medical management, general advice and education, and referral to other services as clinically indicated, according to local practice.
  Arms: Usual Care

SUMMARY:
Chronic musculoskeletal pain is a highly prevalent condition that is often associated with persistent pain, physical disability, and maladaptive psychosocial factors such as pain catastrophizing, fear of movement, and central sensitization. These factors can contribute to pain persistence and reduced quality of life, highlighting the need for multimodal, non-pharmacological interventions that address both physical and psychological dimensions of pain.

The purpose of this study is to evaluate the effectiveness of an active coping program for patients with chronic musculoskeletal pain compared with usual care. The intervention is designed to promote active pain management strategies through education, movement-based exercises, and behavioral approaches aimed at improving pain coping, reducing disability, and addressing psychosocial contributors to chronic pain.

This is a controlled interventional study in which adult patients with chronic musculoskeletal pain will be allocated to either an intervention group receiving the active coping program or a control group receiving usual care. Outcome measures will be assessed at baseline and after completion of the intervention. Primary and secondary outcomes include pain-related disability, pain catastrophizing, fear of movement, symptoms of central sensitization, and health-related quality of life, measured using validated questionnaires.

The findings of this study are expected to provide evidence on the clinical effectiveness of an active coping approach in the management of chronic musculoskeletal pain and to support its implementation in routine clinical practice within primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.

Diagnosis of chronic musculoskeletal pain, defined as pain persisting for more than 3 months.

Ability to understand study procedures and complete self-reported questionnaires.

Ability to participate in an active coping program involving education and movement-based activities.

Provision of written informed consent.

Exclusion Criteria:

* Presence of serious neurological, rheumatologic, or systemic disease that may interfere with participation in the intervention or outcome assessment.

Severe cognitive impairment or psychiatric condition that limits understanding of the study procedures.

Ongoing participation in another structured pain management or rehabilitation program.

Any medical condition that, in the opinion of the investigators, would make participation unsafe or compromise study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | Baseline (Week 0) and post-intervention (Week 8)
  The Pain Catastrophizing Scale (PCS) is a self-reported questionnaire assessing catastrophic thinking related to pain, including rumination, magnification, and helplessness.
  The total score ranges from 0 to 52, with higher scores indicating greater pain catastrophizing (worse outcome).
Roland-Morris Disability Questionnaire (RMDQ) | Baseline (Week 0) and post-intervention (Week 8)
  The Roland-Morris Disability Questionnaire (RMDQ) is a self-reported questionnaire assessing pain-related physical disability in daily activities.
  The total score ranges from 0 to 24, with higher scores indicating greater disability (worse outcome).
Tampa Scale for Kinesiophobia (TSK-11) | Baseline (Week 0) and post-intervention (Week 8)
  The Tampa Scale for Kinesiophobia - 11 item version (TSK-11) is a self-reported questionnaire assessing fear of movement and re-injury related to pain.
  Total scores range from 11 to 44, with higher scores indicating greater kinesiophobia (worse outcome).
Central Sensitization Inventory (CSI) | Baseline (Week 0) and post-intervention (Week 8)
  The Central Sensitization Inventory (CSI) is a self-reported questionnaire used to assess symptoms associated with central sensitization.
  The total score ranges from 0 to 100, with higher scores indicating greater symptom severity related to central sensitization (worse outcome).
36-Item Short Form Health Survey (SF-36) | Baseline (Week 0) and post-intervention (Week 8)
  The 36-Item Short Form Health Survey (SF-36) is a generic self-reported questionnaire assessing health-related quality of life across multiple physical and mental health domains.
  Each domain score ranges from 0 to 100, with higher scores indicating better health-related quality of life (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, Ph.D., Study Director — University of Extremadura
Locations (1):
- University of Extremadura, Badajoz, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No